CLINICAL TRIAL: NCT00000484
Title: Treatment of Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 3
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2000-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Chlorothiazide; Secologanin Tryptamine Alkaloids

INTERVENTIONS:
Drug: chlorothiazide
Drug: Rauwolfia alkaloids

SUMMARY:
To determine whether the long-term treatment of essential hypertension without significant target organ disease materially influenced mortality and/or cardiovascular renal morbidity.

DETAILED DESCRIPTION:
BACKGROUND:

This grant-supported, cooperative, fixed-protocol clinical study was initiated in 1966 and followed a cooperative study of the treatment of renal hypertension initiated in 1960 to evaluate the relative efficacy of several recognized drug regimens for reduction of blood pressure. Six centers (USPHS hospitals) and a coordinating center were involved in the trial.

DESIGN NARRATIVE:

Randomized, double-blind, fixed sample. Three hundred and eighty nine eligible patients were assigned to drug therapy consisting of chlorothiazide plus Rauwolfia serpentina or to placebo.

The study completion date listed in this record was inferred from last publication listed in the Citations section of this study record.

ELIGIBILITY:
Men and women, ages 21-55. Mild essential hypertension (diastolic blood pressure over 90 mm Hg.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1966-04; Study Completion 1979-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Damato — USPHS Hospital; Richard Thurm — USPHS Hospital; Christfried Urner — USPHS Hospital; John Vaillancourt — USPHS Hospital; J. Warbasse — USPHS Hospital; Robert Wells — USPHS Hospital

REFERENCES:
- [Background] U.S. Public Health Service Hospitals Cooperative Study Group. Smith WM, et al: Intervention Trial in Mild Hypertension. Epidemiology and Control of Hypertension. Paul, O (Ed.), Symposia Specialists, Miami, l975, pp. 46l-483.
- [Background] Smith WM. Mild essential hypertension: benefit of treatment: discussion. Ann N Y Acad Sci. 1978 Mar 30;304:74-80. doi: 10.1111/j.1749-6632.1978.tb25573.x. No abstract available. PMID 360933
- [Background] Smith WM, Edlavitch SA, and Krushat WM: U.S. Public Health Service Hospitals Intervention Trial in Mild Hypertension. Hypertension, Determinants, Complications, and Intervention. Onesti G, and Klimt C, (Eds.), Grune & Stratton, New York, l979, pp. 38l-399.
- [Background] Smith WM: Hypertension--Effectiveness of Early Treatment in Preventing Sequellae. Proceedings of the Eisenhower Medical Center. Preventive Interventions in the Practice of Medicine, Spring, l979, pp. 8l-87.
- [Background] Smith WM, Edlavitch SA, and Krushat WM: Prevention of Stroke in Mild Hypertension: Public Health Service Hospitals Trial. Perspectives in Cardiovascular Research, Vol. 4. Prophylactic Approach to Hypertensive Diseases, Yamori Y, Lovenberg W, and Freis ED, (Eds.), Raven Press, New York, l979, pp. 53-62.